CLINICAL TRIAL: NCT04323501
Title: Rehabilitation Treatment and Biomarkers of Post-stroke Recovery: a Pilot Study
Brief Title: Post-stroke Recovery (PSR_e2020)
Acronym: PSR_e2020
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GrantEccellenza_MIUR2020
Record Dates: First submitted 2020-03-12; First posted 2020-03-26 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Stroke
Keywords: Stroke; Self-management; Rehabilitation; Neuronal plasticity; Motivation; Gait; Microbiota; Oxidative stress
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: An experimental pilot study, randomized, controlled and is single-blind, without drug and medical device.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental treatment group (Experimental): This group will undergo an intensive-rehabilitation treatment of post-stroke sensorimotor disability based on a "guided self-rehabilitation contract". This approach is based on the fact that the patient must complete a diary of his self-rehabilitation activity in order to verify its correct and full execution. The treatment protocol will be defined on the basis of the clinical picture (patterns) manifested by the patient (the intensity and frequency of the exercises will be adapted according to the characteristics of each patient). The duration of treatment will be the same for all patients. The exercises will be performed every day throughout the study period (12 months).
  Before undertaking the intensive self-management treatment, each patient will undergo 10 sessions of neurorehabilitation treatment at the UOC Neurorehabilitation of the Integrated University Hospital according to normal clinical practice, during which the patient will be provided with infographic support material.
  Interventions: Other: Experimental treatment
- Control group (Active Comparator): The patients allocated to the control group, during the study period they will undergo conventional outpatient rehabilitation treatment (usual care) at the Neurorehabilitation Unit of the AOUI according to the clinical practice through the procedures provided for by the Health System National.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental treatment — Exercises may include UPPER LIMB Passive exercises (stretching), each one greater or equal to 10 minutes; greater or equal once a day: pectoralis; back muscles and triceps; subscapular muscle; elbow flexor; both pronator muscles; flexor of the wrist and fingers; flexor, adductor and opponent muscles of the thumb.
  Active exercises: multiple repetitions possible in 1 minute each one greater or equal to three times a day: shoulder abduction, flexion, external rotation; elbow extension and supination; wrist extension; finger extension; thumb extension and abduction.
  LOWER LIMB Passive exercises, each one greater or equal to 10 minutes; greater or equal once a day: hamstring; adductor of the hip; gluteus muscles.
  Greater or equal to 5 minutes; greater or equal to twice a day: soleus and gastrocnemius.
  Active exercises: multiple repetitions possible in 1 minute each one greater or equal to three times a day: hip abduction and flexion; knee flexion; dorsiflexion of ankle; seat-standing
  Arms: Experimental treatment group
Other: Control group — Usual care
  Arms: Control group

SUMMARY:
The study presented is part of the departmental project entitled: BEHAVIORS AND WELLNESS: A MULTIDISCIPLINARY APPROACH TO PROMOTE THE QUALITY OF LIFE IN VULNERABILITY CONDITIONS - winner of the MIUR grant "Departments of Excellence", provided by Law 232 of 2016.

The departmental project has the general aim of understanding the interaction between behaviours, motivational and psycho-biological aspects in a situation of neurodegenerative disease and/or mental distress, from which derive six different types of patients that constitute the six lines of research into which the departmental project is divided. The project, as all lines of research, is organized into two essential phases:

* Phase I: the creation of basic models based on the in-depth knowledge of the molecular, structural and functional mechanisms (both physiological and cognitive) as well as on the psychological components (e.g. the ability to cope with the disease and the implementation of strategies functionals to the well-being) which are better indicative of an improvement in the health conditions of the six different patient populations studied;
* Phase II: clinical-applicative integration in which studies will be carried out on the motivations and consequent behaviours in everyday life contexts. Therefore, will be highlighted actions to take place in the healthcare, educational and organizational fields, aimed to promote the implementation of the practices most clearly associated with improving the health conditions highlighted by basic research.

The peculiarity of the studies, that make the departmental project, consists in the effort to encourage translational research, multidisciplinarity and the integration of knowledge, stimulating an innovative dialogue between the different scientific disciplinary sectors present in the department. The purpose is to make evidence-based the whole path related to behaviours and strategies that promote well-being, connecting biological, motivational or behavioural aspects each other, that make it possible to recover or not worsen the conditions of health. The idea is to encourage, where possible, the implementation, even outside or in continuity with the strictly hospital context, of practices aimed at promoting the well-being and quality of life in people in conditions of vulnerability.

Each of the six research lines (1. Young patients with multiple sclerosis; 2. People with chronic brain stroke outcomes; 3. Parkinson's disease patients with symptoms of both physical and mental fatigue; 4. Preschooler population presents "regulatory disturbances"; 5. Migrants seeking international protection; 6. Population in old age and at risk of frailty) is integrated into the purposes and outcome of the departmental project, however, each providing a specific and appropriate study protocol, it is independently submitted to the approval of the Ethics Committee.

DETAILED DESCRIPTION:
Cerebral stroke is the world's second leading cause of death with an incidence of 6.7 million deaths caused each year. Despite the progress made in the prevention and treatment of acute stroke, it remains the main cause of disability in adulthood in industrialized countries with a prevalence of 40% as regards the degrees of disability that significantly affect common daily activities.

Currently, in Italy, the total number of people with long-term disabilities resulting from a stroke has now exceeded one million. However, the rehabilitation pathways of the therapy for the stroke mainly focus on the first weeks/months after the acute event, not always taking into account patient's needs sufficiently in the chronic phase of the disease (> 4-6 months from a stroke). All this is further aggravated by the difficulty of access to treatment and by the reduction in the quality of life, once the hospital phase of taking charge has ended.

The actual organizational model is based on insufficient evidence regarding the mechanisms of post-injury recovery in the subacute and chronic phase of cerebral stroke together with the poor knowledge of the factors related to it and capable of influencing it. This is because the mechanisms able to condition long-term recovery remain unclear, the expression of which can often be interpreted as the reversibility of the functional phenomena of deconditioning / deterioration typical of the chronic phase of the stroke.

In this regard, considering the framework of multidomain disabilities (sensorimotor, cognitive-behavioural, autonomous and psycho-social) that characterizes patients with cerebral stroke, it is necessary to define different factors (clinical-functional, neurophysiological and neuroimaging, genetic-molecular and psychological) which correlates prospectively with the picture of functional recovery and long-term post-stroke disability. All this in order to describe a profile of biomarkers that characterize patients with greater recovery potential, on which to base the development of innovative rehabilitation protocols (based, in particular, on the use of "self-management" programs and innovative technologies) of long term.

STUDY DESIGN This will be an experimental pilot study, without drug or medical device, single-blind randomized controlled trial.

OBJECTIVE OF THE STUDY The general objective is the study of the effects of a protocol innovative rehabilitation based on self-management for the long-term management of the patient with cerebral stroke together with the definition of a profile of clinical-biological, imaging, neurophysiological and genetic/molecular biomarkers related to the effects of this, better defining the post-stroke disability framework. The objectives of the study are related to the research line called "People suffering from chronic stroke outcomes" of the departmental development project entitled "BEHAVIORS AND WELLNESS: A MULTIDISCIPLINARY APPROACH TO PROMOTE THE QUALITY OF LIFE IN VULNERABILITY CONDITIONS".

The study is divided into several Work-packages (WP). In particular, all registered subjects will follow WP1. The other WPs (2 - 7) will be articulated starting from WP1 on the basis of the specific characteristics of each subject included.

OBJECTIVE WP1 As for WP1 (the only interventional WP that defines the main research line), the primary objective is to evaluate the effects of intensive self-management treatment compared to those of "habitual care" on sensory post-stroke sensorimotor disability. The second aspect of WP1 will be: to evaluate the effects of intensive self-management treatment on post-stroke cognitive disability compared to "habitual care"; to evaluate the effects of intensive self-management treatment on post-stroke global disability compared to those of habitual care; evaluate the correlation of structural and functional neuroimaging with the primary outcome (volumetric lesion analysis, lesion site analysis, DTI, fMRI); evaluate the correlation of neurophysiological variables (PEM, PESS, cortical excitability) with the primary outcome.

OBJECTIVE WP2 The main objective of this WP will be to evaluate in patients with ictal damage to different brain regions and investigate complex behavioural functions of fundamental importance for daily life activities. In particular, this WP aims to evaluate cortical plasticity mechanisms through cognitive measures of selective attention (cognitive plasticity) with a view to predicting plasticity in other areas (e.g. motor) in order to guide the planning of rehabilitation protocols more personalized based on the specific characteristics of each patient that take into account the post-stroke multi-domain disability.

OBJECTIVE WP3 The objectives of this WP will be: to explore the characteristics of fatigue (global, physical, mental) in patients suffering from brain stroke outcomes; evaluate markers of the overall health status in patients with brain stroke outcomes; measure the efficiency of walking in patients with brain stroke outcomes.

OBJECTIVE WP4 The goal of this WP is to explore the main psychological characteristics, psychopathology and the presence of psychological distress experienced by patients with stroke and consequent pain. In particular, the idea behind this WP consists in identifying the psychological functioning characteristics typical of the specific pathology on the one hand and the individual aspects on the other, which may have an impact on the rehabilitation process. The usefulness of acting on these aspects could be useful to increase the motivation for neurorehabilitation treatment and its consequent effectiveness.

OBJECTIVE WP5 The objective of this WP is to study changes in the microbiota during disease and after treatment with the aim will be to identify altered bacterial populations. Subsequently, it will be evaluated how lifestyles (movement, psycho-therapeutic approach, etc.) can modify the composition of the microbiota to bring it back to its physiological condition (pre-pathology).

OBJECTIVE WP6 The objective of this WP is to identify a correlation between the expression of miRNA involved in the regulation of neuroplasticity, and prognosis in post-ischemic stroke patients during rehabilitation treatment.

OBJECTIVE WP7 The goal of this WP is the assessment of oxidative stress in the plasma of patients at the onset of the disease and in the rehabilitation recovery phases.

POPULATION Cerebral stroke patients.

The population involved in WP1 will be the starting population from which to derive the population of the other WPs. As for WP 5, 6, 7, the population will follow that of WP1, while the involvement of patients in WP 2, 3, 4 will take place on the basis of further inclusion/exclusion criteria. This means that not all patients enrolled in WP1 will be involved in WP 2, 3, 4.

Enrollment of patients Patients in the sub-acute phase of cerebral stroke (<3 months from the acute event) hospitalized at the UOC Neurorehabilitation of the Integrated University Hospital of Verona (AOUI) will be enrolled. These patients will be offered the opportunity to participate in the study in question, the modalities of which will be presented according to the information document and providing the requested clarifications colloquially. Once informed consent for participation in the study has been obtained, the subject may be subjected to the assessments provided for by WP1 and/or by the other WPs.

Procedures Patients will be enrolled according to the main methods and purposes set out in WP1. Therefore, all enrolled patients will undergo the evaluation and treatment procedures foreseen by WP1. In line with the presence of a post-stroke disability involving multiple domains, subgroups of subjects based on their characteristics can be defined within the sample enrolled for WP1.

LENGHT OF THE STUDY

* First-year - Preparation phase: definition of protocol and WP; presentation of the protocol to the Ethics Committee and its approval; initial acquisition of the devices necessary for carrying out the study and training of the staff for their use.
* Second, third and fourth year - Clinical phase: enrollment, evaluation and treatment of patients; data collection and analysis; progressive acquisition of the devices necessary for carrying out the study and training of the staff for their use; presentation of preliminary results.
* Last year - Final phase: development and implementation of a departmental strategy aimed at integrating the different lines of research developed by the individual areas of intervention; publication of the results obtained.
* Patient involvement: 12 months
* Total duration: 5 years

SAMPLE SIZE Considering as the main outcome measure for WP1 the level of functional impairment measured at the FMA, for which a Minimal Detectable Change value of 5.2 has been defined in the literature, given a level alpha of 5%, a power (beta) of 80% (considering that it is a pilot study) and an SD of 10.2 [28], was calculated that a sample size of 122 total patients (61 for the experimental treatment group and 61 for the control group) may be sufficient to observe any significant difference between the pre and post-treatment conditions. Taking into account a possible drop-out rate of about 10%, the sample size was increased by 12 total subjects (6 for the experimental treatment group and 6 for the control group), reaching a final calculation of 134 patients to enrol.

STATISTICAL ANALYSIS Adequate descriptive statistics will be produced for each WP (1 - 7) (frequency histograms; position or central trend indices: mean, median; variability or sample dispersion indices: standard deviation, interquartile range; construction of confidence intervals) for regarding demographic data and the various variables taken into consideration at each assessment time (see above).

As for WP1, the comparison between the experimental treatment group and the control group subjected to "usual care", with regard to the outcomes considered (FMA and OCS) in the various evaluation times, will be performed through the use of parametric tests ( t-test, ANOVA) or non-parametric (Kruskal Wallis test, Mann-Whitney test) on the basis of data distribution. Correlation and / or regression analyzes will also be performed between neuroimaging data (structural and functional), neurophysiological variables and the main clinical outcome (FMA) at the various assessment times.

With regard to the remaining WPs (2 - 7), the statistical significance of the variations between groups relative to the variables assessed at different times (vide supra) will be assessed through the use of parametric (t-test, ANOVA) or non-parametric tests (Kruskal Wallis test, Mann-Whitney test) based on data distribution. For each variable considered (both longitudinally and transversely) correlation and/or regression analyzes will also be performed with the main clinical outcome (FMA and OCS) of WP1 at the different evaluation times.

Finally, for each WP the statistical significance of the variations with respect to the variables assessed longitudinally intra-group at different times (vide supra) will be assessed through the use of parametric tests (t-test, ANOVA) or non-parametric tests (Friedman test, Wilcoxon test) based on data distribution.

The statistical analysis will be performed using the Statistical Package for Social Science SPSS® version 26.0 software for Macintosh (SPSS Inc., Chicago, IL, USA). For all statistical tests, the significance level is set at 5%.

ELIGIBILITY:
The population involved in work-package (WP) 1 will be the starting population from which to derive the population of the other WPs. As for WP 5, 6, 7, the population will follow that of WP1, while the involvement of patients in WP 2, 3, 4 will take place on the basis of further inclusion/exclusion criteria. This means that not all patients enrolled in WP1 will be involved in WP 2, 3, 4.

WP 1, 5, 6, 7 Inclusion criteria

* Age over 18 years;
* First diagnosis of ischemic brain stroke (ICD9-CM 446, 434) documented radiologically (CT or MRI).
* Presence of post-stroke multidomain disability assessed with Fugl-Meyer assessment (FMA) and with Oxford Cognitive Screen (OCS).
* Patients in the sub-acute phase of cerebral stroke (<3 months from the event) inpatients of the UOC Neurorehabilitation of the Integrated University Hospital of Verona for which the need to continue taking care of post-hospitalization rehabilitation was found.
* The ability of the subject and/or caregiver to understand the instructions provided for the self-management of home disability
* Signature of informed consent

Exclusion criteria

* Contemporary participation in other clinical studies.
* Cognitive impairment defined as a score (corrected) for the Mini-Mental State Examination <23.8.
* Substance abuse.
* Other neurological and orthopaedic pathologies capable of interfering with the study.

Particularly vulnerable populations cannot be included in the study:

* patients with judicial interdiction
* patients for whom a legal guardian has been appointed
* institutionalized patients

Criteria for exit from the study

* Relapse of disease during the study period
* Withdrawal of informed consent to participate in the study
* Impossibility to carry out the assessments foreseen by the study protocol or the rehabilitation treatment according to the defined schedule.

Description of the pathologies studied Outcomes of cerebral stroke with ischemic aetiology (ICD9-CM 446, 434).

WP2 criteria Inclusion criteria

* See inclusion criteria WP 1
* Presence of specific cognitive disorders as assessed by OCS
* Adequate comprehension skills as assessed through the OCS Semantic Test Exclusion criteria
* See exclusion criteria WP 1
* Limited sustained attention span as assessed during the neuropsychological assessment.

WP3 criteria Inclusion criteria

* See inclusion criteria WP 1
* patients suffering from cerebral stroke outcomes in chronic phase (after 3 months from the acute event) or post-hospital discharge
* independent gait or by means of aids (eg cane)
* Adequate comprehension skills as assessed through the OCS Semantic Test Exclusion criteria
* See exclusion criteria WP 1

WP4 criteria Inclusion criteria

* See inclusion criteria WP 1
* Presence of pain following a stroke assessed by Brief Pain Inventory -I
* Adequate understanding and production skills as assessed through OCS language tests Exclusion criteria
* See exclusion criteria WP 1
* Presence of moderate/severe cognitive disorders assessed by OCS which could compromise the insight and communication skills necessary to fill in specific psychological questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the change between the time points on Fugl-Meyer assessment (FMA) | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  The FMA allows quantifying the degree of post-stroke disability through the evaluation of the following 5 domains of interest. In the upper and lower limbs: the motor function; sensory function; the range of motion; joint pain. The last domain is balance control.

SECONDARY OUTCOMES:
Oxford Cognitive Screen (OCS) | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  The Oxford Cognitive Screen is a short and efficient cognitive screening tool that can be delivered at the bedside in acute stroke. OCS is easy to administer and score and importantly is inclusive for patients with aphasia and neglect. OCS returns a single, not divisible visual snapshot of a patient's cognitive profile, which at a glance demonstrates the specific cognitive domain impairments in Attention, Language, Praxis, Number and Memory.
Barthel Index (BI) | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  The Barthel Index explores 10 items related to movement, walking, personal hygiene, ability to eat, intestinal and urinary continence.
  The resulting score expresses the degree of assistance that the patient's condition requires in daily activities. The value zero indicates a totally dependent patient, while the value 100, which represents the maximum, indicates a fully autonomous patient.
Volumetric lesion analysis, lesion site analysis, Diffusion Tensor Imaging DTI, functional Magnetic Resonance Imaging fMRI. | T0 (baseline) - T4 (12 months)
  Correlation of structural and functional neuroimaging with primary outcome measure (volumetric lesion analysis, lesion site analysis, DTI, fMRI)
Motor evoked potentials (MEP), somatosensitive evoked potentials (SSEP) | T0 (baseline) - T4 (12 months)
  Correlation of neurophysiological variables (MEP, SSEP) with the primary outcome.
Transcranial Magnetic Stimulation (TMS) | T0 (baseline) - T2 (6 months)
  Correlation of neurophysiological variables (cortical excitability parameters assessed with TMS) with the primary outcome.

OTHER OUTCOMES:
Outcome measures provided especially for the other work-packages Electroencephalography (EEG) | T0 (baseline) - T2 (6 months)
  Evaluation of physiological measures of cortical activity using electroencephalography. The topography of alpha and beta waves.
Outcome measures provided especially for the other work-packages Electroencephalography (EEG) | T0 (baseline) - T2 (6 months)
  Evaluation of physiological measures of cortical activity using electroencephalography. The latency (ms) of alpha and beta waves.
Outcome measures provided especially for the other work-packages Electroencephalography (EEG) | T0 (baseline) - T2 (6 months)
  Evaluation of physiological measures of cortical activity using electroencephalography. The amplitude (uV) of alpha and beta waves.
Outcome measures provided especially for the other work-packages Multidimensional Fatigue Inventory (MFI) | T2 (6 months)
  The Multidimensional Fatigue Inventory (MFI) aim to measure the frequency and severity of global fatigue (scores from 0 to 100, where higher scores in the MFI scale represent more serious levels of fatigue) and to define the typology of the same (physical or mental), through the analysis of the different scores obtained with the questionnaire.
Outcome measures provided especially for the other work-packages Dual-energy X-ray Absorptiometry (DXA) | T2 (6 months)
  The DXA aim to estimate the following variables: fat mass; lean mass; bone mineral content and total body and regional bone mineral density,
Outcome measures provided especially for the other work-packages Microbiota | T0 (baseline) - T4 (12 months)
  The objective of this work-package is to analyse the microbiota within the first two weeks after stroke and after the treatment (pharmacological and rehabilitative) with the aim to identify the presence of possible different (pre e post) bacterial populations constituting the microbiota. Stool samples will be taken during the hospitalization of stroke patients in the acute phase (<15 days from the event) and subsequently at 12 months.
Outcome measures provided especially for the other work-packages miRNA | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  The levels of expression of specific circulating miRNAs (miR-9, miR-29a-3p, miR-34a, miR-124, miR-146a, miR-223, miR-371-3p, miR-495-3p and miR-941) will be analyzed from serum samples.
Outcome measures provided especially for the other work-packages Biochemistry analysis | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  The level of oxidative stress will be correlated with the severity of the pathology and with the quality and time of recovery of the patient. The following oxidative stress markers will be evaluated on plasma samples: concentration of [GSH] / [GSSG]; concentration of [NO2 -] / [NO3-]; post-translational oxidative modifications of plasma proteins (carbonylation, Tyr-nitration and Cys-glutathionylation).
Outcome measures provided especially for the other work-packages Clinical-psychological evaluation Symptom Checklist-90 scale | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  The Symptom Checklist-90 (SCL-90) is designed to evaluate a broad range of psychological problems and symptoms of psychopathology. It consists of 90 items and takes 12-15 minutes to administer. Each of the 90 items is given a Likert score from 0 (not at all) to 4 (extremely) points, corresponding to the measure of the intensity of the subjective experience of unease. This scale yielding nine scores along primary symptom dimensions and three scores among global distress indices. The primary symptom dimensions that are assessed are somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, and a category of "additional items" which helps clinicians assess other aspects of the client's symptoms.
Outcome measures provided especially for the other work-packages Clinical-psychological evaluation Eysenck Personality Questionnaire-R | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  The Eysenck personality questionnaire - revised is a 100 items self-report questionnaire used to as-sess three dimensions of personality: Neuroticism (emotionality)composed by 24 items, Extraversion by 23 items and Psychoticism(tough-mindedness) with 32 items. It also includes a Lie scale for dissimulation (21items). The response to each item is yes/no.
Outcome measures provided especially for the other work-packages Clinical-psychological evaluation Coping Orientation to Problems Experienced - inventory (COPE-inventory) | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  The Coping Orientation to Problems Experienced - inventory (COPE-inventory) is comprised of 15 four-item scales that assess a variety of coping strategies. Using the dispositional response format, participants indicated how frequently they used each coping strategy on a four-point scale anchored by ''usually do not do this at all'' and ''usually do this a lot''. Each scale total is computed as an unweighted sum of responses to the four items that make up that scale. There is no overall total score.
Outcome measures provided especially for the other work-packages Clinical-psychological evaluation General Self-Efficacy Scale | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  The scale was created to assess a general sense of perceived self-efficacy with the aim in mind to predict coping with daily hassles as well as adaptation after experiencing all kinds of stressful life events. The scale is usually self-administered, as part of a more comprehensive questionnaire. Preferably, the 10 items are mixed at random into a larger pool of items that have the same response format. Time: It requires 4 minutes on average. Scoring: Responses are made on a 4-point scale (1- not at all true; 4- exactly true). Sum up the responses to all 10 items to yield the final composite score with a range from 10 to 40.
Outcome measures provided especially for the other work-packages Clinical-psychological evaluation Acceptance and Action Questionnaire-II scale (AAQ-II scale) | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  The AAQ-II is purported to be a 7-item measure of psychological inflexibility. Participants responded to items using a 7-point Likert scale from 1 (not at all true) to 7 (completely true).
Outcome measures provided especially for the other work-packages Clinical-psychological evaluation Multidimensional Scale of Perceived Social Support | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  It has 12 items divided into three subscales: 4 for family subscale, 4 friends subscale, and 4 significant other subscale. Items were measured on a 5-points.scale from 1 strongly disagree to 5 strongly agree. It provides four scores: one for each subscale and the total.
Outcome measures provided especially for the other work-packages Clinical-psychological evaluation Brief Pain Inventory scale (BPI) | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  The BPI is a patient-completed numeric rating scale that assesses the severity of pain (Severity scale), its impact on daily functioning (Interference scale), and other aspects of pain (e.g., location of pain, relief from medications). Patients are asked to rate separately how their pain interferes with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Total scores on the subscale of pain interference with functions are calculated by adding the scores for each item on pain interference. The four severity and the seven interference items can also each be summed to form composite scores.
Outcome measures provided especially for the other work-packages Clinical-psychological evaluation Stroke Impact Scale (SIS) | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  The current version of the SIS is a 59-item patient-reported outcome measure, covering 8 domains: strength (4 items), hand function (5 items), mobility (9 items), activities of daily living (10 items), memory (7 items), communication (7 items), emotion (9 items), and handicap (8 items). Domains are scored on a metric of 0 to 100, with higher scores indicating better self-reported health.
Outcome measures provided especially for the other work-packages Walking efficiency variables | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  Assessment of the kinematic gait parameters (speed, m/s) by means of video analysis.
Outcome measures provided especially for the other work-packages Walking efficiency variables | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  Assessment of the kinematic gait parameters (amplitude of the step, meters) by means of video analysis.
Outcome measures provided especially for the other work-packages Walking efficiency variables | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  Assessment of the kinematic gait parameters (frequency of the step, number/minute) by means of video analysis.
Outcome measures provided especially for the other work-packages Walking efficiency variables | T0 (baseline) - T1 (3 months) - T2 (6 months) - T3 (9 months) - T4 (12 months)
  Measurement of the energy cost of walking by non-invasive analysis of respiratory exchanges in the mouth (using a portable metabolimeter).

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Smania, MD, Principal Investigator — Universita di Verona; Alessandro Picelli, PhD, Study Director — Universita di Verona
Locations (1):
- Section of Clinical Neurology, Department Neurological, Neuropsychological, Morphological and Movement Sciences, University of Verona, Verona, Italy, Verona, Italy

REFERENCES:
- [Derived] Picelli A, Filippetti M, Del Piccolo L, Schena F, Chelazzi L, Della Libera C, Donadelli M, Donisi V, Fabene PF, Fochi S, Fonte C, Gandolfi M, Gomez-Lira M, Locatelli E, Malerba G, Mariotto S, Milanese C, Patuzzo C, Romanelli MG, Sbarbati A, Tamburin S, Venturelli M, Zamparo P, Carcereri de Prati A, Butturini E, Varalta V, Smania N. Rehabilitation and Biomarkers of Stroke Recovery: Study Protocol for a Randomized Controlled Trial. Front Neurol. 2021 Jan 15;11:618200. doi: 10.3389/fneur.2020.618200. eCollection 2020. PMID 33519698